CLINICAL TRIAL: NCT05848427
Title: The LUSZ COVID-19 Severity Index: A Prognostic and Predictive Score of Mortality for Hospitalized Patients With Covid-19.
Acronym: LUSZ_SCORE
Status: Recruiting | Type: Observational
Sponsor: Lebanese University (Other)
Collaborators: Hospital Saydet Zgharta University Medical Center (Unknown)
Responsible Party: Principal Investigator, Nehman Makdissy, Professor, Lebanese University
Other Study IDs: The COVID-19 LUSZ SCORE
Record Dates: First submitted 2023-05-05; First posted 2023-05-08 (Actual); Last update posted 2024-04-05 (Actual); Status verified 2024-04

CONDITIONS: COVID-19
Keywords: covid-19; SARS-CoV-2; comorbidities; score; inflammation; LUSZ; WHO ordinal severity scale; treatment; IL6; antiviral; antiretroviral; immunosuppressive; antagonist
MeSH Terms: conditions — COVID-19; Inflammation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- LUSZ WOSS-3: hospitalized COVID-19 patients classified as WOSS-3 (as per the WHO Ordinal Severity Scale) who didn't need oxygen therapy
  Interventions: Other: LUSZ P
- LUSZ WOSS-4: hospitalized COVID-19 patients classified as WOSS-4 (as per the WHO Ordinal Severity Scale) who needed oxygen therapy by mask or traditional nasal cannula
  Interventions: Other: LUSZ P
- LUSZ WOSS-5: hospitalized COVID-19 patients classified as WOSS-5 (as per the WHO Ordinal Severity Scale) who needed oxygen therapy NIMV or HFNC
  Interventions: Other: LUSZ P
- LUSZ WOSS-6: hospitalized COVID-19 patients classified as WOSS-6 (as per the WHO Ordinal Severity Scale) who needed oxygen therapy IMV & intubation
  Interventions: Other: LUSZ P

INTERVENTIONS:
Other: LUSZ P — LUSZ protocol applied to WOSS in-hospitalized Covid-19 patients: a Corticosteroid Therapy-enhanced Standard Care (CTSC), a standard care enhanced by corticosteroid (methylprednisolone) treatment.

SUMMARY:
The coronavirus disease 2019 (COVID-19) has spread rapidly and caused a global pandemic, as defined by the WHO, within a short period of time. The prognostic of disease severity is still a challenge and early identification of risk factors to be involved in its progression is of high importance. The scoring of variables related to worse outcomes is key for a targeted and/or advanced protocol. Besides, the need for a predictive-wide model is mandatory for hospitalized unvaccinated patients to avoid any delay in the characterization of severe illness and the development of complications. The LUSZ COVID-19 Severity Index was developed as a predictive tool based on >100 risk factors/biomarkers, that could effectively identify high-risk patients and prevent mortality.

DETAILED DESCRIPTION:
The scientific community is in urgent need of reliable biomarkers related to COVID-19 disease progression, in order to stratify high-risk patients. The rapid disease spread necessitates the immediate categorization of patients into risk groups following diagnosis, to ensure optimal resource allocation. Novel biomarkers are needed to identify patients who will suffer rapid disease progression to severe complications and death. The identification of novel biomarkers is strictly related to the understanding of viral pathogenetic mechanisms, as well as cellular and organ damage. Effective biomarkers would be helpful for screening, clinical management, and prevention of serious complications.

Indeed, previous studies suggested and developed predictive scores (CALL, Chosen, HA2T2, ANDC, ABC2-SPH, ICOP, SEIMC, IRS, NLP, APACHE II, GRAM, and others) that estimate the severity of the disease, the risk of needing invasive mechanical ventilation (IMV) among patients with COVID-19 and the risk of mortality. Many scores including so many relevant parameters have been used to predict the status of a patient. In addition to comorbidities, age, etc., some hematological parameters, including white blood cell (WBC), lymphopenia, c-Reactive Protein (CRP), and some biochemical parameters, such as lactate dehydrogenase (LDH), creatine kinase (CK), and troponin were reported to be associated with COVID-19 severity. In fact, the patient's initial laboratory scoring is useful but not sufficient to avoid mortality: high neutrophil count (>0.7 × 103/μL), lymphopenia (<0.8 × 103/μL), elevated CRP (>4.75 mg/dL), and elevated LDH (>593 U/L) were the most important predictors of mortality. Another prognostic marker the lymphocyte-to-CRP ratio (LCR), was also helpful. A rise in the NLR and a decline in LCR correlates with the severity of COVID-19. Specifically, a low LCR at presentation was seen to predict ICU admission and the need for invasive ventilation. Patients critically ill with COVID-19 had a hyperinflammation, the associated biomarkers may be beneficial for risk stratification. Many studies found other associations with serum CRP, procalcitonin (PCT), D-dimer, and serum ferritin. Subsequent studies demonstrate that the inflammatory response plays a critical role in COVID-19, and inflammatory cytokine storm increases the severity of COVID-19. In fact, the serum levels of IL-6 can effectively assess disease severity and predict outcomes in patients with COVID-19. So, these prognostic models have been introduced to guide treatment and resource management.

In this study, we aimed to specify high-risk factors and biomarkers of fatal outcomes in hospitalized subjects with coronavirus depending on many variables analysis, and also to compare the efficacy of targeted treatments (antiviral, antiretroviral, immunosuppressive antagonist, etc.) in order to help clinicians better choose a therapeutic strategy.

The population had been divided into groups according to the WHO Ordinal Clinical Severity Scale on which the LUSZ SCORE was applied; The percentage of mortality, in and out of the hospital, the length of stay in the hospital, the pulmonary inflammatory lesions and their distribution, the SARS-CoV-2 IgM and IgG variations at admission, the inflammatory markers, the complete blood count, the coagulation factors and enzymes, proteins and electrolytes profile, glucose and lipid profile, and others were measured before and after LUSZ scoring. The establishment of this novel predictive scoring model of disease progression may help identify patients with COVID-19 who may subsequently develop a critical illness. Thus, we can improve the therapeutic effect and reduce the mortality of COVID-19 with more accurate and efficient use of medical resources, which helps to deliver proper treatment according to each case.

ELIGIBILITY:
Inclusion Criteria: (1) admission to hospital, (2) fulfills WHO case definition, including a positive PCR for COVID-19 from any specimen (e.g., nasopharyngeal, throat, saliva, urine, stool, other bodily fluid), (3) not received any therapy (radiotherapy, chemotherapy, corticotherapy, hormonotherapy, immunotherapy, anti-inflammatory, antibiotics, antiparasitic, antiviral, antibacterial, convalescent plasma, monoclonal antibodies, or other treatments such as hydroxychloroquine and azithromycin) before admission and samples' collection, and (4) Spo2 < 90%.

Exclusion Criteria: (1) Non-SARS-CoV-2, (2) active indication and use for one of the investigational products (e.g., HIV positive if antiretroviral agents were used), (3) allergy or hypersensitivity to one of the investigational products (Lopinavir/Ritonavir, Remdesivir, Tocilizumab) or other contraindication, (4) progression to death is imminent and inevitable within the next 24 hours, irrespective of the provision of treatments, (5) received any therapy (radiotherapy, chemotherapy, hormonotherapy, immunotherapy, anti-inflammatory, antibiotics, antiparasitic, antiviral, antibacterial, convalescent plasma, monoclonal antibodies, or other treatments such as hydroxychloroquine and azithromycin) before admission and samples' collection, (6) weight loss during the last 2 years, (7) abdominal surgeries, (8) pregnancy, and (9) SpO2 superior or equal to 90%, and (10) vaccinated individuals were excluded.

-

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: This is a prospective cohort study with data on patients collected and followed up from March 28, 2020, from the SZUMC (as one single medical center; this study will be applied to other centers). All included patients were diagnosed by polymerase chain reaction (PCR) test taken from a nasopharyngeal sample, throat sputum, saliva, urine, stool, or bodily fluid. Analyses were realized upon admission as well 8-10 days after admission. All patients were followed by the principal investigator of the study. The collection of data from each patient in terms of laboratory data, treatments, and outcomes was verified by the principal investigator through the review of clinical records. Selected patients were divided into groups according to the WHO ordinal clinical severity scale.
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2020-03-28 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Survival / Mortality | 1 day to 3 years
  Occurence of survival or death
LOS | up to 3 months
  Time to recovery in-hospital (the length of stay (LOS))
IMV | during the first 3 days of hospitalization
  incidence of mechanical ventilation and incidence of serious adverse effects

SECONDARY OUTCOMES:
Clinical Status | up to 3 years
  Clinical status at days 8-10 by radiology and laboratory assessments

CONTACTS AND LOCATIONS:
Overall Officials: Nehman Makdissy, Professor, Study Chair — Lebanese University
Locations (2):
- Lebanon (2):
  - Lebanese University, Tripoli, Mohafazat Liban-Nord
  - SZUMC, Zghartā, Mohafazat Liban-Nord

IPD SHARING:
Plan to Share IPD: No